CLINICAL TRIAL: NCT03762265
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Oral BTK Inhibitor Rilzabrutinib (PRN1008) in Moderate to Severe Pemphigus
Brief Title: A Study of PRN1008 in Patients With Pemphigus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on lack of efficacy
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17092; PRN1008-012 (Other: Principia Biopharma); 2018-002261-19 (EudraCT Number)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Pemphigus
Keywords: Pemphigus Vulgaris (PV); Pemphigus Foliaceus (PF)
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Then Rilzabrutinib (Placebo Comparator): In BT period, participants received placebo orally twice daily (BID) up to 37 weeks along with sponsor-provided corticosteroids (CS). After at least two weeks of control of disease activity (CDA; no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 milligrams (mg) prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 in OLE period and those who were eligible after OLE period completion, continued the same treatment until Week 109 in LTE period according to protocol-specified criteria.
  Interventions: Drug: Rilzabrutinib; Drug: Placebo
- Rilzabrutinib Then Rilzabrutinib (Experimental): In BT period, participants received rilzabrutinib 400 mg orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 in OLE period and those who were eligible after OLE period completion, continued the same treatment until Week 109 in LTE period according to protocol-specified criteria.
  Interventions: Drug: Rilzabrutinib

INTERVENTIONS:
Drug: Rilzabrutinib — Pharmaceutical form: Tablet Route of administration: Oral
Drug: Placebo — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Placebo Then Rilzabrutinib

SUMMARY:
This was a Phase 3 randomized, parallel-group, double-blind, placebo-controlled trial (blinded treatment [BT] period) followed by an open-label extension [OLE] period intended to evaluate the efficacy and safety of oral PRN1008 in moderate to severe pemphigus. After completing the open-label extension period, eligible participants might continue in a long term extension (LTE) Period of 48 weeks.

DETAILED DESCRIPTION:
A total of 131 male or female participants with newly diagnosed or relapsing moderate to severe pemphigus (pemphigus vulgaris [PV] or pemphigus foliaceus [PF]) were enrolled in the trial worldwide.

The trial would last 68 weeks (approximately 17 months) for each participant. For participants eligible to enroll in the LTE, the trial might last up to 116 weeks.

Participants were randomized at Day 1, using a 1:1 ratio to receive PRN1008 or placebo twice per day, by relapsing/newly diagnosed disease history (newly diagnosed defined as within 6 months of screening).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18 to 80 years old with moderate to severe, newly diagnosed or relapsing PV or PF, with a clinical presentation and histopathology consistent with PV or PF.
* Positive circulating anti-desmoglein 1 (anti-dsg1) or 3 autoantibody titer.
* At screening, pemphigus disease area index score of at least 9 points for relapsing participants or at least 15 points for newly diagnosed participants.
* Adequate hematologic, hepatic, and renal function.
* Effective means of contraception.

Exclusion Criteria:

* Suspected paraneoplastic pemphigus and other forms of pemphigus that were not PV or PF.
* Previous use of a Bruton tyrosine kinase inhibitor.
* Pregnant or lactating women.
* Electrocardiogram clinically significant abnormalities.
* A history of malignancy of any type within 5 years before Day 1, other than surgically excised non-melanoma skin cancers or in situ cervical cancer.
* Use of immunologic response modifiers as concomitant medication and with the washout period.
* Use of proton pump inhibitor drugs such as omeprazole and esomeprazole within 3 days of Day 1.
* Concomitant use of known strong-to-moderate inducers or inhibitors of cytochrome P450 3A (CYP3A) within 3 days or 5 half-lives (whichever is longer) of Day 1
* Use of CYP3A-sensitive substrate drugs.
* Had received any investigational drug within the 30 days before Day 1.
* History of drug abuse within the previous 12 months.
* Alcoholism or excessive alcohol use.
* Any other clinically significant disease, condition or medical history that, in the opinion of the Investigator, would interfere with participant safety, trial evaluations, and/or trial procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (12):
  - Central Recruiting (Principia Biopharma), Boca Raton, Florida
  - Central Recruiting (Principia Biopharma), Coral Gables, Florida
  - Central Recruiting (Principia Biopharma), Atlanta, Georgia
  - Central Recruiting (Principia Biopharma), Ann Arbor, Michigan
  - Central Recruiting (Principia Biopharma), Rochester, Minnesota
  - Central Recruiting (Principia Biopharma), Albuquerque, New Mexico
  - Central Recruiting (Principia Biopharma), New York, New York
  - Central Recruiting (Principia Biopharma), Chapel Hill, North Carolina
  - Central Recruiting (Principia Biopharma), Durham, North Carolina
  - Central Recruiting (Principia Biopharma), Cleveland, Ohio
  - Central Recruiting (Principia Biopharma), Austin, Texas
  - Central Recruiting (Principia Biopharma), Murray, Utah
- Argentina (2):
  - Central Recruiting (Principia Biopharma), Buenos Aires
  - Central Recruiting (Principia Biopharma), San Nicolás
- Australia (3):
  - Central Recruiting (Principia Biopharma), Fremantle, Western Australia
  - Central Recruiting (Principia Biopharma), Melbourne
  - Central Recruiting (Principia Biopharma), Sydney
- Brazil (3):
  - Central Recruiting (Principia Biopharma), Campinas
  - Central Recruiting (Principia Biopharma), Campo Grande
  - Central Recruiting (Principia Biopharma), Ribeirão Preto
- Bulgaria (3):
  - Central Recruiting (Principia Biopharma), Pleven
  - Central Recruiting (Principia Biopharma), Plovdiv
  - Central Recruiting (Principia Biopharma), Sofia
- Central Recruiting (Principia Biopharma), Winnipeg, Manitoba, Canada
- Croatia (2):
  - Central Recruiting (Principia Biopharma), Osijek
  - Central Recruiting (Principia Biopharma), Zagreb
- France (6):
  - Central Recruiting (Principia Biopharma), Bobigny
  - Central Recruiting (Principia Biopharma), Bordeaux
  - Central Recruiting (Principia Biopharma), Lille
  - Central Recruiting (Principia Biopharma), Pierre-Bénite
  - Central Recruiting (Principia Biopharma), Rouen
  - Central Recruiting (Principia Biopharma), Toulouse
- Germany (8):
  - Central Recruiting (Principia Biopharma), Berlin
  - Central Recruiting (Principia Biopharma), Dresden
  - Central Recruiting (Principia Biopharma), Düsseldorf
  - Central Recruiting (Principia Biopharma), Erlangen
  - Central Recruiting (Principia Biopharma), Heidelberg
  - Central Recruiting (Principia Biopharma), Kiel
  - Central Recruiting (Principia Biopharma), Lübeck
  - Central Recruiting (Principia Biopharma), Münster
- Greece (4):
  - Central Recruiting (Principia Biopharma), Athens
  - Central Recruiting (Principia Biopharma), Ioannina
  - Central Recruiting (Principia Biopharma), Larissa
  - Central Recruiting (Principia Biopharma), Thessaloniki
- Israel (4):
  - Central Recruiting (Principia Biopharma), Beersheba
  - Central Recruiting (Principia Biopharma), Haifa
  - Central Recruiting (Principia Biopharma), Ramat Gan
  - Central Recruiting (Principia Biopharma), Tel Aviv
- Italy (8):
  - Central Recruiting (Principia Biopharma), Brescia
  - Central Recruiting (Principia Biopharma), Catania
  - Central Recruiting (Principia Biopharma), Florence
  - Central Recruiting (Principia Biopharma), Milan
  - Central Recruiting (Principia Biopharma), Padua
  - Central Recruiting (Principia Biopharma), Parma
  - Central Recruiting (Principia Biopharma), Rome
  - Central Recruiting (Principia Biopharma), Torino
- Poland (5):
  - Central Recruiting (Principia Biopharma), Gdansk
  - Central Recruiting (Principia Biopharma), Krakow
  - Central Recruiting (Principia Biopharma), Lublin
  - Central Recruiting (Principia Biopharma), Warsaw
  - Central Recruiting (Principia Biopharma), Wroclaw
- Serbia (2):
  - Central Recruiting (Principia Biopharma), Belgrade
  - Central Recruiting (Principia Biopharma), Novi Sad
- Spain (4):
  - Central Recruiting (Principia Biopharma), Barcelona
  - Central Recruiting (Principia Biopharma), Córdoba
  - Central Recruiting (Principia Biopharma), Madrid
  - Central Recruiting (Principia Biopharma), Pamplona
- Taiwan (3):
  - Central Recruiting (Principia Biopharma), Dalin
  - Central Recruiting (Principia Biopharma), Kaohsiung City
  - Central Recruiting (Principia Biopharma), Taipei
- Turkey (Türkiye) (4):
  - Central Recruiting (Principia Biopharma), Fatih
  - Central Recruiting (Principia Biopharma), Istanbul
  - Central Recruiting (Principia Biopharma), Konyaalti
  - Central Recruiting (Principia Biopharma), Merkez
- Ukraine (4):
  - Central Recruiting (Principia Biopharma), Dnipro
  - Central Recruiting (Principia Biopharma), Kyiv
  - Central Recruiting (Principia Biopharma), Lviv
  - Central Recruiting (Principia Biopharma), Zaporizhzhya
- Central Recruiting (Principia Biopharma), London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 88 active sites in 19 countries. A total of 210 participants were screened from 08 January 2019 to 23 October 2020, of whom 79 participants were screen failures, mainly due to not meeting inclusion criteria. A total of 131 participants were enrolled and randomized in the study, consisted of 3 parts: blinded treatment (BT) period (Baseline to Week 37), open-label extension (OLE) period (Week 37 to Week 61) and long term extension (LTE) Period (Week 61 to Week 109).
Pre-assignment Details: Participants with moderate to severe pemphigus (pemphigus vulgaris [PV] and pemphigus foliaceus [PF]) were randomized (1:1 ratio) to receive either rilzabrutinib or placebo in BT period.
Groups:
- Placebo Then Rilzabrutinib: In BT period, participants received placebo orally twice daily (BID) up to 37 weeks along with sponsor-provided corticosteroids (CS). After at least two weeks of control of disease activity (CDA; no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 milligrams (mg) prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 in OLE period and those who were eligible after OLE period completion, continued the same treatment until Week109 in LTE period according to protocol-specified criteria.
- Rilzabrutinib Then Rilzabrutinib: In BT period, participants received rilzabrutinib 400 mg orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 and those who were eligible after OLE period completion, continued the same treatment until Week 109 in LTE period according to protocol-specified criteria.
Period: BT Period: Weeks 1 to 37
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Started | 66 | 65
Completed | 51 | 62
Not Completed | 15 | 3
Not completed — Adverse Event | 7 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Required prohibited medication | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Other | 0 | 1
Period: OLE Period: Weeks 37 to 61
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Started | 51 | 61 (One participant did not enter OLE Period.)
Completed | 35 | 45
Not Completed | 16 | 16
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 3 | 2
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Study terminated by sponsor | 8 | 10
Not completed — Withdrawal by Subject | 3 | 2
Period: LTE Period: Weeks 61 to 109
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Started | 35 | 34 (11 participants did not enter LTE Period.)
Completed | 6 | 6
Not Completed | 29 | 28
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study terminated by sponsor | 28 | 25
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Placebo Then Rilzabrutinib: In BT period, participants received placebo orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 in OLE period and those who were eligible after OLE period completion, continued the same treatment until Week109 in LTE period according to protocol-specified criteria.
- Total: Total of all reporting groups
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib | Total
Number analyzed (Participants) | 66 | 65 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (14.00) | 50.5 (14.11) | 51.7 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 32 | 29 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 52 | 58 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Complete Remission (CR) With a Corticosteroids Dose of Less Than or Equal to (<=) 10 mg/Day From Week 29 to Week 37: Pemphigus Vulgaris Participants in Modified Intent-to-Treat (PV mITT) Population
Description: Complete remission was defined as absence of new and established lesions and was intended to mean "no disease activity" for 2 consecutive weeks, with Pemphigus Disease Area Index (PDAI) activity score =0 and CS dose <=10 mg. PDAI score weighted for number and size of lesions with score of 0 (absent) to 10 given for skin (12 body locations), scalp and mucous membrane showing disease activity (erosions/blisters or new erythema). PDAI total score ranged from 0 to 250 points representing disease activity (120 points for skin activity; 10 points for scalp activity; 120 points for mucosal activity). Higher score indicated more disease activity. In this outcome measure (OM), percentage of participants who achieved CR while on a daily corticosteroids dose of <=10 mg/day were reported.
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on PV mITT which included randomized PV participants who had received at least one dose of study medication and were analyzed according to the treatment they were allocated to at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
percentage of participants | 18.2 | 24.1
Statistical Analysis 1: Comparison: Placebo Then Rilzabrutinib vs Rilzabrutinib Then Rilzabrutinib; P-value and 95% confidence interval (CI) were based on Cochran-Mantel-Haenszel general association test stratified by disease type (PV or PF) and disease history (newly diagnosed [<=6 months prior to screening] or relapsing [diagnosed greater than [>] 6 months prior to screening]); Test type: Superiority; p = 0.4469, Cochran-Mantel-Haenszel; Difference in percentage = 5.73, 95% CI 2-sided [-9.037 to 20.500], Standard Error of Mean 7.535

2. Primary Outcome: Percentage of Participants Who Achieved Complete Remission With a Corticosteroids Dose of <=10 mg/Day From Week 29 to Week 37: Modified Intent-to-Treat (mITT) Population
Description: Complete remission was defined as absence of new and established lesions and was intended to mean "no disease activity" for 2 consecutive weeks, with PDAI activity score =0 and CS dose <=10 mg. PDAI score weighted for number and size of lesions with score of 0 (absent) to 10 given for skin (12 body locations), scalp and mucous membrane showing disease activity (erosions/blisters or new erythema). PDAI total score ranged from 0 to 250 points representing disease activity (120 points for skin activity; 10 points for scalp activity; 120 points for mucosal activity). Higher score indicated more disease activity. In this OM, percentage of participants who achieved CR while on a daily corticosteroids dose of <=10 mg/day were reported.
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on mITT population which included all randomized participants (i.e. PV + PF participants) who had received at least one dose of study medication and were analyzed according to the treatment they were allocated to at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
percentage of participants | 18.2 | 26.2
Statistical Analysis 1: Comparison: Placebo Then Rilzabrutinib vs Rilzabrutinib Then Rilzabrutinib; P-value and 95% CI were based on Cochran-Mantel-Haenszel general association test stratified by disease type (PV or PF) and disease history (newly diagnosed [<=6 months prior to screening] or relapsing [diagnosed >6 months prior to screening]); Test type: Superiority; p = 0.2510, Cochran-Mantel-Haenszel; Difference in percentage = 8.13, 95% CI 2-sided [-5.752 to 22.019], Standard Error of Mean 7.085

3. Secondary Outcome: Cumulative Oral Corticosteroid Dose From Baseline to Week 37: PV mITT Population
Description: The cumulative dose (in milligrams) of sponsor-provided oral CS (prednisone or prednisolone) received by the participants during the BT period was calculated from Baseline to Week 37 and is reported in this OM.
Time Frame: Baseline to Week 37
Population: Analysis was performed on PV mITT population.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
milligrams | 5653.2 (3155.97) | 5131.4 (2623.92)

4. Secondary Outcome: Cumulative Oral Corticosteroid Dose From Baseline to Week 37: mITT Population
Description: as for outcome 3
Time Frame: Baseline to Week 37
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
milligrams | 5392.2 (2993.02) | 4860.2 (2545.32)

5. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Week 37: PV mITT Population
Description: Cumulative duration (in days) of CR post first CS dose of <= 10 mg/day from Baseline to Week 37 was analyzed with a zero-inflated negative binomial model with terms of treatment group and disease history, and an offset based on the number of days on blinded treatment period and were reported in this OM. Complete remission was defined as the absence of new and established lesions and was intended to mean "no disease activity".
Time Frame: Baseline to Week 37
Population: Analysis was performed on PV mITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
days | 34.1 (51.58) | 50.5 (67.10)

6. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Week 37: mITT Population
Description: as for outcome 5
Time Frame: Baseline to Week 37
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
days | 34.0 (54.36) | 54.3 (68.76)

7. Secondary Outcome: Time to First Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Week 37: PV mITT Population
Description: Time to first CR was the time (in days) to achieve CR while on CS dose of <=10 mg/day. Complete remission was defined as the absence of new and established lesions to the "no disease activity". Kaplan-Meier method was used for the analysis.
Time Frame: Baseline to Week 37
Population: Analysis was performed on PV mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
days | 252.0 [150.00 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events. | 197.0 [156.00 to NA] — Upper limit of 95% CI was not estimable due to very low number of participants with events.

8. Secondary Outcome: Time to First Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Week 37: mITT Population
Description: as for outcome 7
Time Frame: Baseline to Week 37
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
days | NA [NA to NA] — Median, upper and lower limit of 95% CI was not estimable due to low number of participants with events. | 197.0 [142.00 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.

9. Secondary Outcome: Percentage of Participants Who Achieved Complete Remission With a Corticosteroids Dose of <=5 mg/Day From Week 29 to Week 37: PV mITT Population
Description: Complete remission was defined as the absence of new and established lesions and was intended to mean "no disease activity". In this OM, percentage of participants who achieved CR while on a daily corticosteroids dose of <=5 mg/day were reported.
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on PV mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
percentage of participants | 10.9 | 24.1

10. Secondary Outcome: Percentage of Participants Who Achieved Complete Remission With a Corticosteroids Dose of <=5 mg/Day From Week 29 to Week 37: mITT Population
Description: as for outcome 9
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
percentage of participants | 12.1 | 26.2

11. Secondary Outcome: Percentage of Participants Who Had Pemphigus Disease Area Index (PDAI) Score <3 With a Corticosteroids Dose <=10 mg/Day From Week 29 to Week 37: PV mITT Population
Description: PDAI is specific cutaneous and mucosal disease activity assessment performed by investigator based on evaluation of lesions in well-defined anatomical locations. The score weighted for the number and size of lesions with score of 0 (absent) to 10 given for skin (12 body locations), scalp and mucous membrane showing disease activity (erosions/blisters or new erythema). Thus, PDAI total activity score ranged from 0 to 250 points representing disease activity (120 points for skin activity; 10 points for scalp activity; 120 points for mucosal activity). Higher score indicated more disease activity. In this OM, participants with PDAI score <3 while on a CS dose of <=10 mg/day were reported.
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on PV mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
percentage of participants | 29.1 | 35.2

12. Secondary Outcome: Percentage of Participants Who Had Pemphigus Disease Area Index Score <3 With a Corticosteroids Dose <=10 mg/Day From Week 29 to Week 37: mITT Population
Description: as for outcome 11
Time Frame: From Week 29 to Week 37
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
percentage of participants | 27.3 | 38.5

13. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Weeks 61 and 109: PV mITT Population
Description: Cumulative duration (in days) of CR post all doses of CS <=10 mg/day during Baseline to Week 61 and Baseline to Week 109 were reported in this OM. Complete remission was defined as the absence of new and established lesions to the "no disease activity".
Time Frame: Baseline to Week 61 and Baseline to Week 109
Population: Analysis was performed on PV mITT population, based on data collected up to database lock for the blinded treatment period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
days
  Baseline to Week 61 | 73.8 (95.35) | 112.2 (120.65)
  Baseline to Week 109 | 102.2 (133.22) | 157.0 (179.71)

14. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Weeks 61 and 109: mITT Population
Description: as for outcome 13
Time Frame: Baseline to Weeks 61 and Baseline to Week 109
Population: Analysis was performed on mITT population, based on data collected up to database lock for the blinded treatment period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
days
  Baseline to Week 61 | 78.1 (98.68) | 120.4 (124.38)
  Baseline to Week 109 | 124.6 (153.76) | 171.6 (186.66)

15. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose = 0 mg/Day From Baseline to Weeks 61 and 109: PV mITT Population
Description: Cumulative duration (in days) of CR post all doses of CS =0 mg/day during Baseline to Week 61 and Baseline to Week 109 were reported in this OM. Complete remission was defined as the absence of new and established lesions to the "no disease activity".
Time Frame: Baseline to Week 61 and Baseline to Week 109
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
days
  Baseline to Week 61 | 13.5 (35.33) | 28.6 (52.33)
  Baseline to Week 109 | 28.4 (77.54) | 60.7 (118.87)

16. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose = 0 mg/Day From Baseline to Weeks 61 and 109: mITT Population
Description: Cumulative duration (in days) of CR post all doses of CS dose = 0 mg/day during Baseline to Week 61 and Baseline to Week 109 were reported in this OM. Complete remission was defined as the absence of new and established lesions to the "no disease activity".
Time Frame: Baseline to Week 61 and Baseline to Week 109
Population: Analysis was performed on mITT population, based on data collected up to database lock for the blinded treatment period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
days
  Baseline to Week 61 | 17.6 (38.56) | 33.5 (55.06)
  Baseline to Week 109 | 49.5 (106.14) | 72.5 (125.60)

17. Secondary Outcome: Glucocorticoid Toxicity Index (GTI) - Cumulative Worsening Score (CWS) and Aggregate Improvement Score (AIS) at Week 37: PV mITT Population
Description: GTI assessed glucocorticoid (GC) related morbidity and GC-sparing ability of other therapies; composed of 2 components: Composite GTI and specific list. Composite GTI had 9 domains and specific list had 23 items (11 domains), used as complementary tool to C-GTI. Composite GTI score:sum of 9 domain-specific scores at each visit and cumulative GTI score:sum of composite GTI scores across each visit. 2 cumulative GTI scores: CWS and AIS at Week 37 reported in this OM. CWS assessed cumulative GC toxicity regardless of whether toxicity had lasting effects/was transient. AIS assessed new therapy effectiveness in decreasing any Baseline GC toxicity over time. CWS composite score range: 0 to 439 and AIS composite score range: -346 to 439. In CWS and AIS, minimum score=least toxicity and maximum score=most toxicity. Least square (LS) mean and standard error (SE) from analysis of covariance model using treatment, disease history as fixed effects and Baseline GTI score and CS dose as covariates.
Time Frame: At Week 37
Population: Analysis was performed on PV mITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
units on a scale
  CWS | 54.46 (8.136) | 73.60 (7.397)
  AIS | 9.42 (6.516) | 19.95 (5.924)

18. Secondary Outcome: Glucocorticoid Toxicity Index - Cumulative Worsening Score and Aggregate Improvement Score at Week 37: mITT Population
Description: GTI assessed GC related morbidity and GC-sparing ability of other therapies; composed of 2 components: Composite GTI and specific list. Composite GTI contained 9 domains and specific list contained of 23 items (11 domains), used as complementary tool to C-GTI. Composite GTI score: sum of 9 domain-specific scores at each visit and cumulative GTI score: sum of composite GTI scores across each visit. Two cumulative GTI scores: CWS and AIS at Week 37 were reported in this OM. CWS assessed cumulative GC toxicity regardless of whether toxicity had lasting effects/was transient. AIS assessed new therapy effectiveness in decreasing any Baseline GC toxicity over time. CWS composite score ranged from 0 to 439 and AIS composite score ranged from -346 to 439. For CWS and AIS, minimum score = least toxicity and maximum score = most toxicity. LS mean and SE from analysis of covariance model using treatment, disease history as fixed effects and Baseline GTI score and CS dose as covariates.
Time Frame: At Week 37
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
units on a scale
  CWS | 51.68 (7.368) | 68.15 (6.732)
  AIS | 8.63 (5.730) | 18.23 (5.236)

19. Secondary Outcome: Change From Baseline in Pemphigus Disease Area Index Score at Weeks 5, 13, 25, 37, 61, and 109: PV mITT Population
Description: PDAI is specific cutaneous and mucosal disease activity assessment performed by investigator based on evaluation of lesions in well-defined anatomical locations. The score weighted for the number and size of lesions with score of 0 (absent) to 10 given for skin (12 body locations), scalp and mucous membrane showing disease activity (erosions/blisters or new erythema). Thus, PDAI total activity score ranged from 0 to 250 points representing disease activity (120 points for skin activity; 10 points for scalp activity; 120 points for mucosal activity). Higher score indicated more disease activity. PDAI activity score was measured independently of the CS dose administered in the participants.
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: Analysis was performed on PV mITT population, based on data collected up to database lock for the blinded treatment period. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
units on a scale
  Week 5: number analyzed (Participants) | 52 | 51
  Week 5 | -7.567 (12.6310) | -7.224 (6.9832)
  Week 13: number analyzed (Participants) | 50 | 53
  Week 13 | -11.076 (11.4549) | -13.925 (10.1497)
  Week 25: number analyzed (Participants) | 45 | 50
  Week 25 | -11.333 (13.8064) | -15.292 (10.5552)
  Week 37: number analyzed (Participants) | 41 | 51
  Week 37 | -13.000 (10.9202) | -14.167 (9.8679)
  Week 61: number analyzed (Participants) | 18 | 28
  Week 61 | -12.900 (6.6418) | -16.475 (10.1585)
  Week 109: number analyzed (Participants) | 1 | 2
  Week 109 | -21.300 | -18.250 (9.8288)

20. Secondary Outcome: Change From Baseline in Pemphigus Disease Area Index Score at Weeks 5, 13, 25, 37, 61, and 109: mITT Population
Description: as for outcome 19
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: Analysis was performed on mITT population, based on data collected up to database lock for the blinded treatment period. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
units on a scale
  Week 5: number analyzed (Participants) | 63 | 62
  Week 5 | -7.870 (12.5361) | -7.161 (6.5918)
  Week 13: number analyzed (Participants) | 59 | 64
  Week 13 | -11.253 (12.1328) | -13.139 (10.3317)
  Week 25: number analyzed (Participants) | 54 | 61
  Week 25 | -11.722 (13.2580) | -14.174 (11.1997)
  Week 37: number analyzed (Participants) | 50 | 62
  Week 37 | -12.918 (11.0260) | -13.442 (10.2669)
  Week 61: number analyzed (Participants) | 27 | 39
  Week 61 | -13.793 (8.9794) | -14.649 (11.4991)
  Week 109: number analyzed (Participants) | 3 | 2
  Week 109 | -23.967 (16.4628) | -18.250 (9.8288)

21. Secondary Outcome: Change From Baseline in Autoimmune Bullous Disease Quality of Life (ABQOL) Score at Weeks 5, 13, 25, 37, 61, and 109: PV mITT Population
Description: ABQOL, a 17-item questionnaire is a valid and reliable tool to assess quality of life in participants with autoimmune blistering diseases. Each question score ranged from 0 to 3 points, 0 = never, 1 = occasionally, 2 = sometimes and 3 = all the time, where higher score = poor QOL. The total ABQoL score was calculated by summing the score of each question and it ranged from 0 to 51, where higher score = more QOL impairment.
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: Analysis was performed on PV mITT population, based on data collected up to database lock for the blinded treatment period. Here, 'overall number of participants analyzed'=participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 52 | 51
score on a scale
  Week 5: number analyzed (Participants) | 49 | 49
  Week 5 | -2.20 (6.856) | -4.47 (7.668)
  Week 13: number analyzed (Participants) | 46 | 50
  Week 13 | -4.04 (6.831) | -6.22 (7.218)
  Week 25: number analyzed (Participants) | 43 | 47
  Week 25 | -5.88 (7.443) | -8.32 (7.647)
  Week 37: number analyzed (Participants) | 38 | 47
  Week 37 | -4.53 (7.518) | -7.19 (8.187)
  Week 61: number analyzed (Participants) | 17 | 25
  Week 61 | -7.76 (6.389) | -8.64 (10.140)
  Week 109: number analyzed (Participants) | 1 | 2
  Week 109 | -19.00 | -19.50 (6.364)

22. Secondary Outcome: Change From Baseline in Autoimmune Bullous Disease Quality of Life Score at Weeks 5, 13, 25, 37, 61, and 109: mITT Population
Description: as for outcome 21
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: Analysis was performed on mITT population, based on data collected up to database lock for the blinded treatment period. Here, 'overall number of participants analyzed'=participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 63 | 62
score on a scale
  Week 5: number analyzed (Participants) | 59 | 60
  Week 5 | -2.02 (6.474) | -4.50 (7.324)
  Week 13: number analyzed (Participants) | 56 | 60
  Week 13 | -3.18 (7.262) | -5.93 (7.168)
  Week 25: number analyzed (Participants) | 52 | 58
  Week 25 | -5.23 (7.259) | -7.57 (7.667)
  Week 37: number analyzed (Participants) | 47 | 58
  Week 37 | -4.43 (7.150) | -7.00 (7.843)
  Week 61: number analyzed (Participants) | 25 | 36
  Week 61 | -7.40 (7.416) | -7.47 (9.263)
  Week 109: number analyzed (Participants) | 3 | 2
  Week 109 | -13.00 (6.000) | -19.50 (6.364)

23. Secondary Outcome: Percentage of Participants With Autoimmune Bullous Disease Quality of Life Score of Zero at Weeks 5, 13, 25, 37, 61, and 109: PV mITT Population
Description: ABQOL, a 17-item questionnaire is a valid and reliable tool to assess quality of life in participants with autoimmune blistering diseases. Each question score ranged from 0 to 3 points, 0 = never, 1 = occasionally, 2 = sometimes and 3 = all the time, where higher score = poor QOL. The total ABQoL score was calculated by summing the score of each question and it ranged from 0 to 51, where higher score = more QOL impairment. Percentage of participants with ABQOL score of '0' were reported in this outcome measure.
Time Frame: At Weeks 5, 13, 25, 37, 61, and 109
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
percentage of participants
  Week 5: number analyzed (Participants) | 51 | 49
  Week 5 | 0.0 | 2.0
  Week 13: number analyzed (Participants) | 47 | 50
  Week 13 | 2.1 | 4.0
  Week 25: number analyzed (Participants) | 45 | 48
  Week 25 | 4.4 | 4.2
  Week 37: number analyzed (Participants) | 38 | 48
  Week 37 | 7.9 | 4.2
  Week 61: number analyzed (Participants) | 17 | 25
  Week 61 | 11.8 | 12.0
  Week 109: number analyzed (Participants) | 1 | 2
  Week 109 | 0.0 | 50.0

24. Secondary Outcome: Percentage of Participants With Autoimmune Bullous Disease Quality of Life Score of Zero at Weeks 5, 13, 25, 37, 61, and 109: mITT Population
Description: as for outcome 23
Time Frame: At Weeks 5, 13, 25, 37, 61, and 109
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Groups:
- Rilzabrutinib Then Rilzabrutinib: along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 in OLE period and those who were eligible after OLE period completion, continued the same treatment until Week109 in LTE period according to protocol-specified criteria.
  In BT period, participants received rilzabrutinib 400 mg orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 and those who were eligible after OLE period completion, continued the same treatment until Week 109 in LTE period according to protocol-specified criteria.
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
percentage of participants
  Week 5: number analyzed (Participants) | 61 | 60
  Week 5 | 0.0 | 1.7
  Week 13: number analyzed (Participants) | 57 | 60
  Week 13 | 1.8 | 5.0
  Week 25: number analyzed (Participants) | 54 | 59
  Week 25 | 3.7 | 6.8
  Week 37: number analyzed (Participants) | 47 | 59
  Week 37 | 6.4 | 5.1
  Week 61: number analyzed (Participants) | 25 | 36
  Week 61 | 12.0 | 8.3
  Week 109: number analyzed (Participants) | 3 | 2
  Week 109 | 33.3 | 50.0

25. Secondary Outcome: Change From Baseline in the European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) Score: Visual Analogue Scale (VAS) Scores at Weeks 5, 13, 25, 37, 61, and 109
Description: EQ-5D-5L: standardized measure of health status that provides general assessment of health and wellbeing. EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS scale ranging from 0 to 100, where 0=worst imaginable health state and 100=best imaginable health state, where higher states indicated better outcomes.
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: For this OM, the planned data collection and analysis was not performed because of early termination of the study.
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Change From Baseline in the European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels Score: Individual Dimension at Weeks 5, 13, 25, 37, 61, and 109
Description: EQ-5D-5L: standardized measure of health status that provides general assessment of health and wellbeing. The EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has a 5-level response: no problems, slight problems, moderate problems, severe problems, and extreme problems. Response options are measured with a 5-point Likert scale (for the 5L version). The 5D-5L systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state and lower score indicate worse health state.
Time Frame: Baseline, Weeks 5, 13, 25, 37, 61, and 109
Population: For this OM, the planned data collection and analysis was not performed because of early termination of the study.
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Time to First Complete Remission With a Corticosteroids Dose <=10 mg/Day From Baseline to Weeks 61 and 109
Description: Time to first CR was the time (in days) to achieve CR while on a CS dose of <=10 mg/day from Baseline to Week 61 and from Baseline to Week 109. Complete remission was defined as absence of new and established lesions to the "no disease activity".
Time Frame: Baseline to Week 61 and Baseline to Week 109
Population: For this OM, the planned data collection and analysis was not performed because of early termination of the study.
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Total Number of Disease Relapses/Flares From Initial Control of Disease Activity (CDA) to Week 37: PV mITT Population
Description: Total Number of Disease Relapses/Flares which occurred from initial CDA to Week 37 were reported. CDA was defined as disappearance of new lesions cease to form and established lesions begin to heal. Relapse/flare was defined by the appearance of 3 or more new lesions after CDA and within a month that do not heal spontaneously within 1 week, or by the extension of established lesions, in a participant who had achieved CDA.
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: Analysis was performed on PV mITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 51 | 53
relapses | 0.6 (0.96) | 0.3 (0.55)

29. Secondary Outcome: Total Number of Disease Relapses/Flares From Initial Control of Disease Activity to Week 37: mITT Population
Description: as for outcome 28
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 62 | 64
relapses | 0.6 (0.94) | 0.3 (0.54)

30. Secondary Outcome: Time to Initial Relapse/Flare From Initial Control of Disease Activity to Week 37: PV mITT Population
Description: Time duration (in days) from the time of initial relapse/flare which occurred from initial CDA up to Week 37 were reported in this OM. CDA was defined as the visit at which new lesions cease to form and established lesions begin to heal. Relapse/flare was defined by the appearance of 3 or more new lesions after CDA and within a month that do not heal spontaneously within 1 week, or by the extension of established lesions, in a participant who had achieved CDA. Kaplan-Meier method was used for the analysis.
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 51 | 53
days | 243.0 [144.00 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with the events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of participants with the events.

31. Secondary Outcome: Time to Initial Relapse/Flare From Initial Control of Disease Activity to Week 37: mITT Population
Description: as for outcome 30
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: as for outcome 29
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 62 | 64
days | 243.0 [148.00 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with the events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of participants with the events.

32. Secondary Outcome: Percentage of Participants With 3 or More New Lesions Within 1 Month That do Not Heal Spontaneously Within 1 Week, or With Extension of Established Lesions at Week 37: PV mITT Population
Description: Percentage of Participants With 3 or More New Lesions Within past 1 month that do not heal spontaneously within past 1 week, or with extension of established lesions, were assessed at Week 37 and reported in this OM.
Time Frame: At Week 37
Population: Analysis was performed on PV mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 55 | 54
percentage of participants | 58.2 | 35.2

33. Secondary Outcome: Percentage of Participants With 3 or More New Lesions Within 1 Month That do Not Heal Spontaneously Within 1 Week, or With Extension of Established Lesions at Week 37: mITT Population
Description: as for outcome 32
Time Frame: At Week 37
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65
percentage of participants | 59.1 | 36.9

34. Secondary Outcome: Percentage of Participants With at Least One Disease Relapse/Flare From Initial Control of Disease Activity to Week 37: PV mITT Population
Description: CDA was defined as the visit at which new lesions cease to form and established lesions begin to heal. Disease relapse/flare was defined by the appearance of 3 or more new lesions after CDA and within a month that do not heal spontaneously within 1 week, or by the extension of established lesions, in a participant who had achieved CDA. Percentages were calculated based on number of participants assessed (i.e. participants achieved CDA) in each treatment group. Percentage of participants with at least one disease relapse/flare from Initial CDA to Week 37 were reported in this OM.
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: Analysis was performed on PV mITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 51 | 53
percentage of participants | 43.1 | 28.3

35. Secondary Outcome: Percentage of Participants With at Least One Disease Relapse/Flare From Initial Control of Disease Activity to Week 37: mITT Population
Description: as for outcome 34
Time Frame: From initial CDA up to Week 37 (i.e., during any time from Baseline up to Week 37)
Population: as for outcome 29
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 62 | 64
percentage of participants | 43.5 | 29.7

36. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Week 37 to Week 61: PV mITT Population
Description: Cumulative duration (in days) of CR post first dose of CS <=10 mg/day from Week 37 to Week 61 were reported in this OM. Complete remission was defined as the absence of new and established lesions and was intended to mean "no disease activity".
Time Frame: From Week 37 to Week 61
Population: Analysis was performed on PV mITT population, based on data collected up to database lock for the blinded treatment period. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 42 | 50
days | 52.0 (59.01) | 62.5 (67.59)

37. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose <=10 mg/Day From Week 37 to Week 61: mITT Population
Description: as for outcome 36
Time Frame: From Week 37 to Week 61
Population: Analysis was performed on mITT population, based on data collected up to database lock for the blinded treatment period. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 51 | 61
days | 57.1 (59.99) | 67.1 (68.03)

38. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose = 0 mg/Day From Week 37 to Week 61: PV mITT Population
Description: Cumulative duration (in days) of CR post first dose of CS = 0 mg/day from Week 37 to Week 61 were reported in this OM. Complete remission was defined as the absence of new and established lesions and was intended to mean "no disease activity".
Time Frame: From Week 37 to Week 61
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 42 | 50
days | 17.7 (39.60) | 30.5 (53.92)

39. Secondary Outcome: Cumulative Duration of Complete Remission With a Corticosteroids Dose = 0 mg/Day From Week 37 to Week 61: mITT Population
Description: as for outcome 38
Time Frame: From Week 37 to Week 61
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Then Rilzabrutinib | Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 51 | 61
days | 22.8 (42.58) | 35.3 (56.32)

40. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and does not necessarily had to have a causal relationship with the treatment. Serious AEs (SAEs) were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were the AEs that developed or worsened or became serious after the administration of first dose of study drug in each period.
Time Frame: BT Period: From Day 1 of Week 1 to Week 37, OLE Period: from Week 37 to Week 61 and LTE Period: from Week 61 up to 4 weeks after the last dose at Week 109 (i.e., up to Week 113)
Population: Analysis was performed on safety population which included all participants who had received at least one dose of study medication and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- BT Period: Placebo: Participants received placebo orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37.
- BT Period: Rilzabrutinib: Participants received rilzabrutinib 400 mg orally BID up to 37 weeks along with Sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone per day from Week 29 to Week 37.
- OLE Period: Placebo Then Rilzabrutinib: Eligible participants post completion of BT period (after receiving placebo), entered OLE period and received rilzabrutinib 400 mg orally BID up to Week 61 in OLE period.
- OLE Period: Rilzabrutinib Then Rilzabrutinib: Eligible participants post completion of BT period (after receiving rilzabrutinib), entered OLE period and received rilzabrutinib 400 mg orally BID up to Week 61 in OLE period.
- LTE Period: Placebo Then Rilzabrutinib; LTE Period: Rilzabrutinib Then Rilzabrutinib: Eligible participants post completion of OLE period (after receiving rilzabrutinib), entered LTE period and continued to receive rilzabrutinib 400 mg BID until Week 109 in LTE period.
Arm/Group | BT Period: Placebo | BT Period: Rilzabrutinib | OLE Period: Placebo Then Rilzabrutinib | OLE Period: Rilzabrutinib Then Rilzabrutinib | LTE Period: Placebo Then Rilzabrutinib | LTE Period: Rilzabrutinib Then Rilzabrutinib
Number analyzed (Participants) | 66 | 65 | 51 | 61 | 35 | 34
Participants
  TEAE | 54 | 55 | 33 | 35 | 18 | 14
  TESAE | 10 | 6 | 4 | 0 | 1 | 2

41. Secondary Outcome: Pharmacokinetics (PK): Plasma Concentration of Rilzabrutinib
Description: Data for this OM was not planned to be collected and analyzed for placebo arm of the study.
Time Frame: Pre-dose and 2 hours post-dose on Day 1
Population: Analysis was performed on PK population which included all participants who had received at least one dose of study medication and had sufficient data for PK analysis.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Groups:
- Rilzabrutinib: In BT period, participants received rilzabrutinib 400 mg orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37. Post completion of BT period, eligible participants received rilzabrutinib 400 mg BID up to Week 61 and those who were eligible after OLE period completion, continued the same treatment until Week 109 in LTE period according to protocol-specified criteria.
Arm/Group | Rilzabrutinib
Number analyzed (Participants) | 65
nanograms per milliliter
  Day 1: pre-dose | NA (NA) — Pre-dose concentration was below limit of quantification (0.1 nanogram per milliliter) and thus mean and standard deviation data were not calculable.
  Day 1: 2-hour post-dose | 273.13 (264.136)

42. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Antibody Levels - Anti-desmoglein 1 (Anti-dsg 1) and Anti-desmoglein 3 (Anti-dsg 3) at Weeks 13, 25, 37, 49, 61, 73, 85, 97, and 109: PV mITT Population
Description: Anti-dsg1 and anti-dsg3 autoantibody levels was assessed by enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Baseline, Weeks 13, 25, 37, 49, 61, 73, 85, 97, and 109
Population: Analysis was performed on PV mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units/milliliter
Groups:
- Placebo: In BT period, participants received placebo orally BID up to 37 weeks along with sponsor-provided CS. After at least two weeks of CDA (no new lesions and established lesions begin to heal), based on protocol-specified clinical criteria, investigators could decrease the CS dose to a minimum of 5 mg prednisone/prednisolone per day from Week 29 to Week 37.
Arm/Group | Placebo | Rilzabrutinib
Number analyzed (Participants) | 55 | 54
units/milliliter
  Baseline: Anti-dsg1 | 108.4 (288.97) | 85.9 (139.17)
  Baseline: Anti-dsg3 | 392.5 (697.52) | 464.1 (668.22)
  Change at Week 13: Anti-dsg1: number analyzed (Participants) | 48 | 52
  Change at Week 13: Anti-dsg1 | 60.6 (116.32) | 15.4 (34.20)
  Change at Week 13: Anti-dsg3: number analyzed (Participants) | 48 | 52
  Change at Week 13: Anti-dsg3 | 197.1 (320.37) | 99.8 (146.65)
  Change at Week 25: Anti-dsg1: number analyzed (Participants) | 45 | 46
  Change at Week 25: Anti-dsg1 | 48.2 (93.15) | 17.5 (37.44)
  Change at Week 25: Anti-dsg3: number analyzed (Participants) | 45 | 46
  Change at Week 25: Anti-dsg3 | 218.6 (314.74) | 153.7 (351.56)
  Change at Week 37: Anti-dsg1: number analyzed (Participants) | 41 | 47
  Change at Week 37: Anti-dsg1 | 42.0 (95.02) | 24.1 (60.01)
  Change at Week 37: Anti-dsg3: number analyzed (Participants) | 41 | 47
  Change at Week 37: Anti-dsg3 | 204.4 (313.26) | 213.9 (389.85)
  Change at Week 49: Anti-dsg1: number analyzed (Participants) | 28 | 39
  Change at Week 49: Anti-dsg1 | 12.1 (18.66) | 17.1 (31.99)
  Change at Week 49: Anti-dsg3: number analyzed (Participants) | 28 | 39
  Change at Week 49: Anti-dsg3 | 215.6 (327.22) | 277.1 (575.77)
  Change at Week 61: Anti-dsg1: number analyzed (Participants) | 17 | 27
  Change at Week 61: Anti-dsg1 | 12.0 (20.61) | 12.5 (26.08)
  Change at Week 61: Anti-dsg3: number analyzed (Participants) | 17 | 27
  Change at Week 61: Anti-dsg3 | 252.3 (439.45) | 223.5 (271.69)
  Change at Week 73: Anti-dsg1: number analyzed (Participants) | 16 | 17
  Change at Week 73: Anti-dsg1 | 12.8 (23.21) | 10.5 (26.34)
  Change at Week 73: Anti-dsg3: number analyzed (Participants) | 16 | 17
  Change at Week 73: Anti-dsg3 | 237.1 (412.33) | 157.6 (186.82)
  Change at Week 85: Anti-dsg1: number analyzed (Participants) | 11 | 11
  Change at Week 85: Anti-dsg1 | 11.7 (24.31) | 14.2 (28.05)
  Change at Week 85: Anti-dsg3: number analyzed (Participants) | 11 | 11
  Change at Week 85: Anti-dsg3 | 169.9 (349.29) | 132.4 (189.76)
  Change at Week 97: Anti-dsg1: number analyzed (Participants) | 5 | 7
  Change at Week 97: Anti-dsg1 | 3.6 (5.27) | 4.7 (8.60)
  Change at Week 97: Anti-dsg3: number analyzed (Participants) | 5 | 7
  Change at Week 97: Anti-dsg3 | 193.0 (330.12) | 95.4 (180.66)
  Change at Week 109: Anti-dsg1: number analyzed (Participants) | 1 | 2
  Change at Week 109: Anti-dsg1 | 1.0 | 2.0 (0.0)
  Change at Week 109: Anti-dsg3: number analyzed (Participants) | 1 | 2
  Change at Week 109: Anti-dsg3 | 0.0 | 94.0 (115.97)

43. Secondary Outcome: Pharmacodynamics: Change From Baseline in Antibody Levels - Anti-desmoglein 1 (Anti-dsg 1) and Anti-desmoglein 3 (Anti-dsg 3) at Weeks 13, 25, 37, 49, 61, 73, 85, 97 and 109: mITT Population
Description: Anti-dsg1 and anti-dsg3 autoantibody levels was assessed by ELISA method.
Time Frame: Baseline, Weeks 13, 25, 37, 49, 61, 73, 85, 97, and 109
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units/milliliter
Arm/Group | Placebo | Rilzabrutinib
Number analyzed (Participants) | 66 | 65
units/milliliter
  Baseline: Anti-dsg1 | 132.2 (275.92) | 141.7 (366.74)
  Baseline: Anti-dsg3 | 328.8 (651.84) | 385.8 (632.71)
  Change at Week 13: Anti-dsg1: number analyzed (Participants) | 57 | 63
  Change at Week 13: Anti-dsg1 | 73.7 (116.08) | 39.8 (102.35)
  Change at Week 13: Anti-dsg3: number analyzed (Participants) | 57 | 63
  Change at Week 13: Anti-dsg3 | 166.1 (302.25) | 82.5 (138.29)
  Change at Week 25: Anti-dsg1: number analyzed (Participants) | 54 | 57
  Change at Week 25: Anti-dsg1 | 65.6 (105.99) | 40.5 (106.10)
  Change at Week 25: Anti-dsg3: number analyzed (Participants) | 54 | 57
  Change at Week 25: Anti-dsg3 | 182.4 (298.18) | 124.3 (320.96)
  Change at Week 37: Anti-dsg1: number analyzed (Participants) | 50 | 57
  Change at Week 37: Anti-dsg1 | 59.5 (101.58) | 37.0 (68.28)
  Change at Week 37: Anti-dsg3: number analyzed (Participants) | 50 | 57
  Change at Week 37: Anti-dsg3 | 167.8 (293.78) | 176.5 (362.67)
  Change at Week 49: Anti-dsg1: number analyzed (Participants) | 37 | 50
  Change at Week 49: Anti-dsg1 | 31.9 (53.27) | 44.1 (102.07)
  Change at Week 49: Anti-dsg3: number analyzed (Participants) | 37 | 50
  Change at Week 49: Anti-dsg3 | 163.4 (298.38) | 216.4 (520.01)
  Change at Week 61: Anti-dsg1: number analyzed (Participants) | 26 | 38
  Change at Week 61: Anti-dsg1 | 41.5 (68.66) | 44.6 (88.74)
  Change at Week 61: Anti-dsg3: number analyzed (Participants) | 26 | 38
  Change at Week 61: Anti-dsg3 | 165.3 (372.10) | 159.2 (249.62)
  Change at Week 73: Anti-dsg1: number analyzed (Participants) | 23 | 24
  Change at Week 73: Anti-dsg1 | 43.5 (87.58) | 48.5 (139.91)
  Change at Week 73: Anti-dsg3: number analyzed (Participants) | 23 | 24
  Change at Week 73: Anti-dsg3 | 165.2 (358.15) | 112.0 (171.90)
  Change at Week 85: Anti-dsg1: number analyzed (Participants) | 16 | 15
  Change at Week 85: Anti-dsg1 | 22.3 (39.62) | 42.1 (105.90)
  Change at Week 85: Anti-dsg3: number analyzed (Participants) | 16 | 15
  Change at Week 85: Anti-dsg3 | 116.9 (296.51) | 97.9 (170.97)
  Change at Week 97: Anti-dsg1: number analyzed (Participants) | 9 | 9
  Change at Week 97: Anti-dsg1 | 21.9 (46.36) | 52.2 (141.86)
  Change at Week 97: Anti-dsg3: number analyzed (Participants) | 9 | 9
  Change at Week 97: Anti-dsg3 | 107.6 (254.47) | 76.0 (161.13)
  Change at Week 109: Anti-dsg1: number analyzed (Participants) | 3 | 2
  Change at Week 109: Anti-dsg1 | 4.7 (4.73) | 2.0 (0.00)
  Change at Week 109: Anti-dsg3: number analyzed (Participants) | 3 | 2
  Change at Week 109: Anti-dsg3 | 1.0 (1.73) | 94.0 (115.97)

ADVERSE EVENTS:
Time Frame: BT Period: From Day 1 of Week 1 to Week 37, OLE Period: from Week 37 to Week 61 and LTE Period: from Week 61 up to 4 weeks after the last dose at Week 109 (i.e., up to Week 113)
Description: Reported AEs and deaths were TEAEs that developed/worsened in grade or became serious after the administration of first dose of study drug in each period. Analysis was performed on safety population. For the OLE and LTE period, AE data for individual arms as well as for the combined population were analyzed and reported under the respective arm.
Groups:
- OLE Period: Overall (All Participants): All eligible participants post completion of BT period (after receiving placebo/rilzabrutinib), entered OLE period and received rilzabrutinib 400 mg orally BID up to Week 61 in OLE period.
- LTE Period: Overall (All Participants): All eligible participants post completion of OLE period (after receiving rilzabrutinib), entered LTE period and continued to receive rilzabrutinib 400 mg BID until Week 109 in LTE period.
Arm/Group | BT Period: Placebo | BT Period: Rilzabrutinib | OLE Period: Placebo Then Rilzabrutinib | OLE Period: Rilzabrutinib Then Rilzabrutinib | OLE Period: Overall (All Participants) | LTE Period: Placebo Then Rilzabrutinib | LTE Period: Rilzabrutinib Then Rilzabrutinib | LTE Period: Overall (All Participants)
All-Cause Mortality (participants affected / at risk) | 2/66 | 0/65 | 0/51 | 0/61 | 0/112 | 0/35 | 0/34 | 0/69
Serious Adverse Events (participants affected / at risk) | 10/66 | 6/65 | 4/51 | 0/61 | 4/112 | 1/35 | 2/34 | 3/69
Other Adverse Events (participants affected / at risk) | 41/66 | 47/65 | 18/51 | 22/61 | 40/112 | 11/35 | 7/34 | 18/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT Period: Placebo (N=66) | BT Period: Rilzabrutinib (N=65) | OLE Period: Placebo Then Rilzabrutinib (N=51) | OLE Period: Rilzabrutinib Then Rilzabrutinib (N=61) | OLE Period: Overall (All Participants) (N=112) | LTE Period: Placebo Then Rilzabrutinib (N=35) | LTE Period: Rilzabrutinib Then Rilzabrutinib (N=34) | LTE Period: Overall (All Participants) (N=69)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Steroid Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vogt-Koyanagi-Harada Disease (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism Arterial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pemphigus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BT Period: Placebo (N=66) | BT Period: Rilzabrutinib (N=65) | OLE Period: Placebo Then Rilzabrutinib (N=51) | OLE Period: Rilzabrutinib Then Rilzabrutinib (N=61) | OLE Period: Overall (All Participants) (N=112) | LTE Period: Placebo Then Rilzabrutinib (N=35) | LTE Period: Rilzabrutinib Then Rilzabrutinib (N=34) | LTE Period: Overall (All Participants) (N=69)
Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (4)
Oral Herpes (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Tinea Versicolour (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 7 (8) | 16 (17) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 6 (7) | 11 (14) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 12 (14) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 9 (14) | 2 (2) | 3 (5) | 5 (7) | 1 (1) | 1 (1) | 2 (2)
Vision Blurred (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (8) | 5 (6) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (7) | 4 (6) | 3 (5) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 8 (9) | 4 (4) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (12) | 8 (8) | 2 (2) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (10) | 1 (1) | 2 (3) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Skin Striae (Skin and subcutaneous tissue disorders) | 1 (4) | 6 (8) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (4) | 5 (6) | 0 (0) | 1 (1) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 10 (11) | 15 (16) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 4 (7) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated prematurely by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03762265/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03762265/SAP_001.pdf